CLINICAL TRIAL: NCT06368830
Title: Characterizing Oral and Swallowing Function in Older Adults Presenting to the Emergency Department
Brief Title: Oral and Swallowing Function in Older Adults
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0337; A534100 (Other: UW Madison); Protocol Version 10/22/25 (Other: UW Madison)
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Oropharyngeal Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples will be retained and human DNA sequences will not be collected from the saliva samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 3-ounce water swallow test — Bedside water swallow dysphagia screen where vocal quality of the participant is assessed before and after swallowing 3 ounces of water
Diagnostic Test: Kayser-Jones Brief Oral Health Status Examination (BOHSE) — Scored assessment of the lymph nodes, lips, tongue, tissue inside of cheek, floor and roof of mouth, gums between teeth and/or under artificial teeth, saliva, condition of natural/artificial teeth, chewing position of teeth, and oral cleanliness
Diagnostic Test: Tongue pressure — Maximum isometric lingual pressure at the front and back of tongue will be measured by placing an air-filled pressure bulb on the surface of the oral tongue and having participants press the bulb "as hard as possible" against the hard palate
Diagnostic Test: Test of Masticating and Swallowing Solids (TOMASS) — Measurement of bites, masticatory cycles, swallows, and time taken to consume a cracker
Diagnostic Test: Respiratory function tests — Participants will take a maximum inhalation and forcefully exhale into a spirometer to measure maximum expiratory pressure (MEP), fully exhale their air and take a maximal inhalation into the spirometer to measure maximum inspiratory pressure (MIP), and produce a single strong cough into to spirometer to measure peak expiratory flow (PEF) and forced expiratory volume (FEV1)

SUMMARY:
The purpose of this study is to learn about oral and swallowing function in older adults presenting to the emergency department. The hypothesis is that older adults often have problems with oral and swallowing function and these problems relate to other conditions. Study activities are done during the emergency department visit and include providing saliva samples, completing a bedside water swallow test, completing oral function assessments, completing respiratory function tests, and answering survey questions.

DETAILED DESCRIPTION:
Oropharyngeal dysphagia is characterized by changes in swallow event timing, biomechanics, and pressure generation that occur with advancing age resulting in aspiration of bacteria-laden saliva, food, and liquid into the lungs. Currently, oral and swallowing function is not routinely or comprehensively assessed in older adults despite poor oral health and oropharyngeal dysphagia being known risk factors for pneumonia, the leading infectious cause of mortality among adults 65+. This study seeks to extensively characterize oral and swallowing function in older adults presenting to the emergency department to clarify the relationship of oral hypofunction, dysphagia, and the upper airway microbiome. To achieve this aim, study procedures include a bedside dysphagia screen, oral health assessment, tongue pressure measurement, masticatory function assessment, respiratory function tests, salivary compositional analysis, oral microbiome analysis, and microphysiological system analysis which applies saliva samples to a bronchiolar lumen model to mimic aspiration and quantify cellular and tissue responses to the saliva microbiome and secreted mediators.

Per amendment approved 10/29/2025: Saliva samples for microbiota analysis will not be collected from participants enrolled after 10/22/2025.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60
* Clinically stable and able (not NPO) to safely drink water and eat a saltine cracker per ED provider

Exclusion Criteria:

* Prisoner
* Non-English speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older adults presenting to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Positive oropharyngeal dysphagia screen prevalence | During emergency department visit, approximately 2-5 minutes for bedside dysphagia screen and 5-10 minutes for patient reported swallowing function
  Number of participants with positive oropharyngeal dysphagia screen identified through bedside dysphagia screen and patient reported swallowing function

SECONDARY OUTCOMES:
Mean brief oral health status examination (BOHSE) score | During emergency department visit, approximately 2-5 minutes
  Score 0 - 20 with 20 indicating the worst oral health
Oral dryness prevalence | During emergency department visit, up to 10 minutes for saliva collection
  Number of participants with stimulated salivary flow rate (volume saliva/collection time) less than two standard deviations below published norms
Decreased tongue pressure prevalence | During emergency department visit, approximately 2-5 minutes
  Number of participants with maximum isometric lingual pressures at front or back tongue location less than fifth percentile for published age-matched norms
Decreased masticatory function prevalence | During emergency department visit, approximately 2-5 minutes
  Number of participants with test of masticating and swallowing solids (TOMASS) greater than two standard deviations above published age- and sex-matched norms for any of four components: number of bites, number of masticatory cycles, number of swallows, total time
pH of saliva sample | During emergency department visit, up to 10 minutes for saliva collection
  pH 0-14 of saliva as measured by digital pH meter
Extensional viscosity of saliva sample | During emergency department visit, up to 10 minutes for saliva collection
  Extensional viscosity of saliva as measured by an extensional rheometer
Salivary Substance P Concentration | During emergency department visit, up to 10 minutes for saliva collection
  Protein concentration (ng/mL) of Substance P in saliva
Oral microbiome | During emergency department visit, up to 10 minutes for saliva collection
  Comparison of microbial community composition in buccal mucosa, tongue dorsum, and saliva based on oral and swallowing function
Cell barrier function | During emergency department visit, up to 10 minutes for saliva collection
  Diffusion assays to quantify cell barrier function in bronchiole and blood vessel model after application of saliva to bronchiolar lumen
Protein composition | During emergency department visit, up to 10 minutes for saliva collection
  Multiplex bead-based ELISA to identify concentration (ng/mL) of proteins in bronchiole and blood vessel model after application of saliva to bronchiolar lumen
Gene expression | During emergency department visit, up to 10 minutes for saliva collection
  Quantification of gene expression in bronchiole and blood vessel model after application of saliva to bronchiolar lumen
Immunofluorescent staining | During emergency department visit, up to 10 minutes for saliva collection
  Quantification of immunofluorescent staining in bronchiole and blood vessel model after application of saliva to bronchiolar lumen
Immune cell trafficking | During emergency department visit, up to 10 minutes for saliva collection
  Quantification of immune cell trafficking in bronchiole and blood vessel model after application of saliva to bronchiolar lumen

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Pulia, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the study will be shared after deidentification to researchers whose proposed use of the data has been approved by principal investigator Dr. Michael Pulia.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months after publication of primary outcomes and ending 5 years after that date.
Access Criteria: Proposals should be directed to Dr. Michael Pulia at mpulia-lab@medicine.wisc.edu. If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.